CLINICAL TRIAL: NCT00583570
Title: Phosphorus Improvement Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Responsible Party: Ashwini Sehgal MD, MetroHealth Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB06-01323; IRB06-01323
Record Dates: First submitted 2007-12-20; First posted 2007-12-31 (Estimated); Last update posted 2009-04-01 (Estimated); Status verified 2009-03

CONDITIONS: Hyperphosphatemia
MeSH Terms: conditions — Hyperphosphatemia | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Behavioral: dietary education

INTERVENTIONS:
Behavioral: dietary education — dietary education

SUMMARY:
Specific Aim: To determine the effect of a phosphorus additives educational intervention on serum phosphorus levels.

Hypothesis: Educating dialysis patients regarding phosphate containing additives will result in improved serum phosphorus levels.

DETAILED DESCRIPTION:
The amount of phosphorus in the American diet has increased considerably, primarily from phosphorus-containing additives in convenience and ready to eat foods (Calvo 1996). It is estimated that, depending on individual food choices, additives add as much 1000 mg/day of phosphorus to the diet (Bell). Phosphorus in additives is almost entirely absorbed while only 60% of naturally occurring phosphorus is absorbed (Uribarri 2003). Education regarding high phosphorus foods is a key component of hyperphosphatemia management (Ford 2004, Cupisti 2004), but the use of phosphorus additives may make it difficult for patients and dietitians to estimate phosphorus content of foods. It has been suggested that hyperphosphatemia is a nutritional barrier to preventing renal bone disease and that an intervention focusing on phosphate containing food additives has great potential (Sherman). Our objective is to determine the effect of an educational intervention regarding phosphate additives on serum phosphorus about 300 chronic hemodialysis patients at Centers for Dialysis Care (CDC) and Fresenius Medical Care (FMC) in Cuyahoga County. Facilities will be randomized to intervention and control groups. All dietitians and eligible patients at the intervention facilities will be invited to take part in the intervention. All dietitians and consenting eligible patients at control facilities will form a usual care group. Prior to the trial, demographic and medical characteristics, lab data and medications will be collected for the previous three months using a chart abstraction and patient interview form. Demographic characteristics include age, sex, race, education and insurance status. Medical characteristics include dialysis dose, binder prescription, vitamin D dosing, cause of renal failure, number of months on dialysis, and major co-morbid conditions. Lab data will include albumin, calcium, phosphorus, serum bicarbonate, and PTH. Medication data will include binder prescription and bone medications. In the first month of the trial study coordinators will meet with intervention and control subjects and assess basic knowledge regarding phosphorus content of foods and label reading. Intervention subjects will also receive education regarding phosphorus additives and their effect on the phosphorus content of foods, a laminated card listing common phosphorus additives, and a handout about additives in foods from fast food restaurants where they eat. The subject will be instructed to use the materials when shopping or eating out to avoid phosphorous additives. During the 2nd month of the trial, study coordinators will contact intervention subjects by phone to reinforce educational materials and answer questions. Control subjects will be contacted and asked about shopping and eating habits. During the 3rd month the interviews from month 1 will be repeated for both intervention and control subjects to assess changes in knowledge. Intervention subjects will also be asked to evaluate the phosphorus additives tool and provide feedback for evaluating the ease of use and utility. Having a control group that receives attention but not the key intervention (phosphorus containing additives education and tools) will allow us to distinguish the effect of attention from the effect of the intervention. Chart abstraction data on labs, dialysis dose, binder prescription, and vitamin D dosing will be collected for all three months of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Most recent phosphorus and mean phosphorus over last 3 months > 5.5 mg/dL
* Age ≥ 18 years
* On chronic hemodialysis ≥ 6 months
* English speaking

Exclusion Criteria:

* Mentally incompetent
* AIDS
* Cancer
* Terminal illness
* Pregnancy
* Nursing home residence
* No telephone access
* In another phosphorus related study
* Unable to identify written words

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2007-05; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
To determine the effect of a phosphorus additives educational intervention on serum phosphorus levels. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ashwini Sehgal, MD, Principal Investigator — MetroHealth Medical Center

REFERENCES:
- [Result] Sullivan C, Sayre SS, Leon JB, Machekano R, Love TE, Porter D, Marbury M, Sehgal AR. Effect of food additives on hyperphosphatemia among patients with end-stage renal disease: a randomized controlled trial. JAMA. 2009 Feb 11;301(6):629-35. doi: 10.1001/jama.2009.96. PMID 19211470
- [Derived] Campbell ZC, Dawson JK, Kirkendall SM, McCaffery KJ, Jansen J, Campbell KL, Lee VW, Webster AC. Interventions for improving health literacy in people with chronic kidney disease. Cochrane Database Syst Rev. 2022 Dec 6;12(12):CD012026. doi: 10.1002/14651858.CD012026.pub2. PMID 36472416